CLINICAL TRIAL: NCT05174156
Title: Study on the Biomarker of First-line Immunotherapy Combined With Chemotherapy in Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Nanjing Geneseeq Technology Inc. (Industry); Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-IO-BIO-1
Record Dates: First submitted 2021-12-15; First posted 2021-12-30 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Advanced Esophageal Cancer
MeSH Terms: interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biomarker study and treatment study (Experimental): All enrolled patients undergo biomarker study and treatment study.
  * Biomarker study: the baseline tumor tissue will be collected and analyzed via NGS and mIHC
  * Treatment study: SHR-1210 plus albumin-bound paclitaxel and platinum-based chemotherapy
  Interventions: Drug: Combination therapy

INTERVENTIONS:
Drug: Combination therapy — SHR-1210 (camrelizumab) + albumin-bound paclitaxel + Carboplatin

SUMMARY:
This study intends to explore the predictive biomarkers by Next-generation sequencing (NGS) and multiple immunohistochemistry (mIHC) for the treatment of SHR-1210 in combination with paclitaxel and platinum in advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable locally advanced/ recurrent or distant metastatic esophageal squamous cell carcinoma confirmed by histology or cytology;
* Not received any previous systematic antitumor therapy.
* Eastern Cooperative Oncology Group (ECOG) fitness status score was 0 or 1 within 3 days before the first administration of the intervention.
* 8-10 tumor tissue samples can be provided.
* Demonstrate good organ and bone marrow function.
* Consent to participate in the contraceptive methods related to clinical research.

Exclusion Criteria:

* Have a history of allergy to monoclonal antibodies, any component of SHR-1210, albumin-paclitaxel, carboplatin, and other platinum drugs;
* Weight loss > 20% in the past 3 months.
* Major surgery within 28 days prior to enrollment.
* Have received systemic chemotherapy or radiation therapy for esophageal cancer.
* Had a myocardial infarction within the past 6 months.
* Have any medical history or current evidence, treatment, or laboratory abnormalities that prevent the subject from participating fully in the study with the investigator's opinion.
* Prior treatment with immunotherapy drugs.
* Received live vaccine within 30 days prior to initial administration of the investigational drug.
* Have been diagnosed with immunodeficiency or are receiving immunosuppressive treatment.
* Another malignancy is known to exist.
* Have active infections that require systemic treatment.
* Pregnant or lactating, or planning to become pregnant or become a father during the study period (180 days for lactating subjects receiving carboplatin) from the beginning of the screening visit until 120 days after the last dose of the study intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to approximately 1 year
  ORR is determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 1 year
  It is defined as the time from enrollment to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment.
Overall Survival (OS) | up to approximately 1 year
  Defined as the time from the enrollment to death from any cause
Disease Control Rate (DCR) | up to approximately 1 year
  The proportion of patients who have achieved complete response， partial response and Stable disease assessed by investigators according to Recist v 1.1.
Adverse events (AEs) | up to approximately 1 year
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE v 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided